CLINICAL TRIAL: NCT01228916
Title: Community-Partnered Tobacco Control in Underserved Dominican Republic Communities
Brief Title: Community-Partnered Dominican Republic Tobacco Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Deborah Ossip, Principal Investigator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01CA132950-01A2 (NIH)
Record Dates: First submitted 2010-10-25; First posted 2010-10-27 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Tobacco Use Cessation; Second Hand Tobacco Smoke
Keywords: tobacco; smoking; secondhand smoke
MeSH Terms: conditions — Tobacco Use Cessation; Smoking | interventions — Tobacco Use Cessation Devices; Tobacco Smoke Pollution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tobacco Cessation and Secondhand Smoke Reduction (Experimental): Community based interventions to raise awareness regarding secondhand smoke exposure, clean indoor air laws, smokefree homes, risks of tobacco use and benefits of cessation; include talks, healthcare provider training, radio public service announcements and talk shows, tleevision interviews, cessation classes and individual sessions, health fairs, community marches for smokefree spaces, materials and resources for assisting in tobacco use cessation, estsablishing smokefree homes, adhering to smokefree laws
  Interventions: Behavioral: Tobacco Cessation and Secondhand Smoke Reduction
- Delayed Intervention Control (No Intervention): Assessment only during comparison period (no interventions will be provided over and above any secular trends in communities); delayed intervention will be provided at end of 1 year comparison period

INTERVENTIONS:
Behavioral: Tobacco Cessation and Secondhand Smoke Reduction — Awareness raising and resources for cessation and secondhand smoke reduction
  Other Names: tobacco cessation; secondhand smoke; smokefree homes
  Arms: Tobacco Cessation and Secondhand Smoke Reduction

SUMMARY:
Tobacco use and tobacco-caused illnesses and death are increasing in developing countries globally, so it is critical to study these countries in order to effectively address the tobacco epidemic. The proposed project will test the effectiveness of community-based interventions for secondhand smoke and quitting smoking in eight underserved communities in the Dominican Republic. The project will also partner with communities and national and international groups to determine whether the methods and interventions from this study in the Dominican Republic can also be used to help other countries in the region and underserved groups in the United States.

DETAILED DESCRIPTION:
The globalization of the tobacco epidemic poses significant morbidity and mortality burdens, with the brunt of impact increasingly borne by low-middle income countries. Research partnerships between investigators from high-income countries with well developed tobacco control research programs and their counterparts in low-middle income countries are needed to effectively address this global public health crisis. The Dominican Republic (DR) is a key site that mirrors the trends in Latin America: it is a low-middle income tobacco growing country with significant tobacco use and high levels of secondhand smoke exposure, and it is at a very early stage of tobacco control. The proposed project will assess baseline knowledge, attitudes, exposures, and behaviors regarding tobacco use and secondhand smoke, provide a randomized controlled trial of community-partnered interventions around secondhand smoke and tobacco cessation, and develop and implement a dissemination plan for national and regional impact and translation of methods and results to other underserved groups as appropriate. A multimethod assessment approach will be used, to include qualitative community assessments (RAPs), a series of quantitative surveys (household surveillances, community and smoker cohort surveys, and health care provider surveys), and a biomarker assessment of secondhand smoke exposure. Eight economically disadvantaged communities will be randomized to intervention or control conditions in a lagged treatment design; interventions will be developed and implemented based on the evidence base from other countries and from a current DR trial, and on input from national and local DR workgroups using a community partnered approach. The intervention is hypothesized to decrease tobacco use rates, increase the number of smokefree homes, denormalize smoking, increase awareness of and change attitudes regarding tobacco use and secondhand smoke risks, decrease exposure to secondhand smoke, and increase health care provider intervention in intervention- relative to control communities, with differences by geographic and demographic characteristics to be examined. The project will also engage international, national, and local DR workgroups to maintain communication of findings to key partners, host a national DR tobacco control conference with regional representation, and develop other action steps for local and regional dissemination of findings and evidence based interventions, resources, and infrastructures. Finally, the project will coordinate with the University of Rochester Clinical and Translational Sciences Institute for translation of current evidence based approaches and methodologies for implementation in the DR, and to explore whether any methodologies or interventions from the proposed trial in the DR can be translated to underserved groups in the United States. Effectively engaging early stage low-middle income countries in tobacco control research will be critical to reducing tobacco use and the burden of tobacco-caused illnesses globally.

ELIGIBILITY:
Inclusion Criteria: For main study: adults (age 18 and older), speak and understand Spanish. For biomarker sub-study (hair samples): children 10 years or younger.

Exclusion Criteria: Non-Spanish speaker, younger than 18 years (except for biomarker sub-study), anyone with questionable capacity or clear decisional impairment.

-

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3273 (Actual)
Dates: Start 2010-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Self-Reported Tobacco Use | Yrs 5
  Self report of current use of any tobacco product

SECONDARY OUTCOMES:
Self Reported Exposure to Secondhand Smoke | Yrs 5
  Home smoking policies, implementation of clean indoor air laws, frequency of being close enough to breathe someone else's smoke
Self-Reported Tobacco Use | Year 4
  Self-reported use of any tobacco products after one year intervention-control period and prior to replication of intervention in control communities.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J Ossip, PhD, Principal Investigator — University of Rochester
Locations (1):
- Centro de Atencion Primaria Juan XXIII, Santiago de los Caballeros, Dominican Republic, Dominican Republic